CLINICAL TRIAL: NCT06670131
Title: Neck Pain in Ukrainian Higher Education Students: Epidemiology and Risk Factors
Brief Title: This Observational Study, Which is Being Implemented by Obtaining Statistical Data From a Google-form Filled Out by Students of Ukrainian Higher Education Institutions, Aims to Investigate the Epidemiological Features of Neck Pain and Possible Risk Factors
Status: Not yet recruiting | Type: Observational
Sponsor: Ukrainian Medical Stomatological Academy (Other)
Responsible Party: Sponsor
Other Study IDs: 22324012024
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Cervicalgia; Neck Pain
Keywords: neck pain; students; risk factors
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to analyze the epidemiological, demographic, social, behavioural and neuropsychological factors of neck pain in students of higher medical education institutions in Ukraine.

To achieve the aim of this study, we will conduct an anonymous survey among medical students seeking master's degrees in Ukrainian higher education institutions.

The questionnaire will be distributed among the student community in special chats and groups in messengers.

DETAILED DESCRIPTION:
The study aims to analyze the epidemiological, demographic, social, behavioural, and neuropsychological factors of neck pain in students of higher medical education institutions in Ukraine.

To achieve the planned study's goal, an anonymous survey of students seeking higher education in the field of knowledge 22-Health care of Ukrainian higher education institutions will be conducted.

The study is planned to do the following:

1. To assess the prevalence and severity of neck pain among students of higher medical education in Ukrainian higher education institutions.
2. To study the limitations of vital activity of higher education students in Ukrainian higher education institutions due to neck pain.
3. To investigate the level of anxiety, depression and stress in neck pain in higher education students of Ukrainian higher education institutions.
4. To study the duration and quality of sleep in higher education students of Ukrainian higher education institutions in the presence of neck pain.
5. To identify and analyze the prevalence of neck pain among students of higher medical education in Ukrainian higher education institutions.
6. To identify the dependence of neck pain intensity on the time of self-study (preparation for classes);
7. To identify the relationship between the intensity of neck pain and the duration of use of electronic devices with a static forward head tilt;
8. To identify the relationship between the intensity of neck pain and the level of perceived stress;
9. To analyze the demographic, social, behavioural and psychological risk factors for neck pain in students of higher medical education in Ukrainian higher education institutions.
10. To develop a program of educational activities for the correction and prevention of neck pain among medical students.

The student survey will be conducted using the Google Forms service.

The survey form contains questions formulated by the researchers and blocks of questions formulated following several instruments:

* Neck Disability Index (NDI);
* Generalized Anxiety Disorder scale (GAD-7);
* The Patient Health Questionnaire (PHQ-9);
* Perceived Stress Scale (PSS-10);
* Social Support Scale (SSS);
* Pittsburgh Sleep Quality Index (PSQI). Given the absence of a validated Ukrainian version of the Social Support Questionnaire, its components will be used in the structure of the questionnaire in the author's translation and internal consistency will be calculated using Cronbach's alpha criterion based on the data of a pilot study with 50 respondents.

The questionnaire will be distributed among the student community in special chats and groups in messengers.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* the presence of injuries, inflammatory and hereditary diseases of the spine
* inadequate answers to open questions:
* sleep duration more than 24 hours
* sleep duration less than 1 hour
* duration of stay with head tilted forward during the day more than 24 hours
* height less than 100 cm and more than 220 cm;
* weight less than 40 kg and more than 150 kg;
* identical answers to all questions of the questionnaire - all A, all B, etc.

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: An anonymous survey of students - higher education students in the field of knowledge 22 - Health care of Ukrainian higher education institutions will be conducted
Sampling Method: Non-Probability Sample
Enrollment: 441 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Neck pain disability index (NDI) | 12.2024-02.2026
  Information about how neck pain has affected ability to cope with everyday life.
GAD-7 Anxiety | 12.2024-02.2026
  Screening tool and severity measure for generalised anxiety disorder
Depression Questionnaire (PHQ-9) | 12.2024-02.2026
  Since the questionnaire relies on patient self-report, all responses should be verified by the clinician, and a definitive diagnosis is made on clinical grounds taking into account how well the patient understood the questionnaire, as well as other relevant information from the patient.
Perceived Stress Scale (PSS-10) | 12.2024-02.2026
  Stress levels will be assessed.
Social Support Scale (SSS) | 12.2024-02.2026
  The Social Support Scale (SSS) is an instrument that can be used to measure a person's availability of perceived social support.
Pittsburgh Sleep Quality Index (PSQI) | 12.2024-02.2026
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval.